CLINICAL TRIAL: NCT03045458
Title: Associations of Alveolar Bone Loss, Clinical Parameters and Interleukin-1β Levels in One and Two Stage Surgical Procedures: A Randomized Prospective Trial
Brief Title: Associations of Alveolar Bone Loss and Interleukin-1β Levels in One and Two Stage Surgical Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Collaborators: Dicle University (Other)
Responsible Party: Principal Investigator, Tuba Talo yıldırım, assistant professor, Firat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D.Ü.D.F.E.K.2010/02
Record Dates: First submitted 2017-01-25; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Implant Infection; Alveolar Bone Loss
Keywords: one stage dental implant; two stage dental implant; Interleukin-1β
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Dental Implants

STUDY DESIGN:
Intervention Model Description: In the surgical operations, 20 tissue-level and 20 bone-level dental implants 12 mm in length and 4.8 mm in diameter were inserted in Group I and Group II, respectively.
Masking Description: Only the surgeon knows detail about the groups of participants. Participant, care provider,outcomes assessor have no knowledge of groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Tissue level dental implant (Active Comparator): Tissue level dental implants (Straumann AG, Waldenburg, Switzerland) were inserted in patients group I (n=20).
  Interventions: Device: tissue level dental implant
- Bone level dental implant (Active Comparator): Bone level dental implants (Straumann AG, Waldenburg, Switzerland ) were inserted in patients group II (n=20).
  Interventions: Device: Bone level dental implant

INTERVENTIONS:
Device: tissue level dental implant — After local anesthesia, full thickness flaps were reflected, and osteotomies were prepared in the first mandibular molar sites. In these surgical operations, 20 tissue-level implants 12 mm in length and 4.8 mm in diameter were inserted in Group I. Cover screw was removed and replaced with healing abutments.
  Other Names: Straumann AG, Waldenburg, Switzerland, dental implant
  Arms: Tissue level dental implant
Device: Bone level dental implant — After local anesthesia, full thickness flaps were reflected, and osteotomies were prepared in the first mandibular molar sites. In these surgical operations, 20 bone-level dental implants 12 mm in length and 4.8 mm in diameter were inserted inGroup II. Three months later, second-stage surgery was performed and implant exposed into the oral cavity. Cover screw was removed and replaced with healing abutments. Three months waited for second surgery in bone level implants.
  Other Names: Straumann AG, Waldenburg, Switzerland, dental implant
  Arms: Bone level dental implant

SUMMARY:
The present study was compared the level of alveolar bone loss, clinical parameters and IL-1β in PICF in one- or two-stage surgical procedures. Half of the patients were performed tissue level implant while other half were performed bone level implant.

DETAILED DESCRIPTION:
The present study included 40 healthy patients (24 males and 16 females; mean age, 30.75 ± 8.58 years) who had one tooth absent in the mandible, at the Department of Periodontology, Dicle University, Diyarbakir, Turkey, between 2010 and 2011. All patients were informed in detail about the study protocol, and they were asked to sign informed consent forms. Ethics committee approval was obtained from Dicle University Ethics Committee for this study (D.Ü.D.F.E.K.2010/02)

This study was designed as a prospective, randomized, controlled study. Randomization was performed prior to surgery by opening a sequentially numbered sealed envelope corresponding to the patient recruitment number. Investigators received randomization instructions only after enrolling a subject and immediately prior to surgery. The participants were randomly divided into two groups. A one-stage surgical procedure was performed on 20 patients (Group I) and a two-stage surgical procedure was performed on the other 20 patients (Group II). The primary outcome of the study was a change in alveolar bone level at the implant site between T0 and T2 months after surgery measured on CBCT. The secondary outcomes between T0, T1, and T2 were changes the level of IL-1β PICF, probing pocket depth (PPD), modified plaque index (mPI), modified gingival index (mGI), and modified bleeding index (mBI). All implants (Straumann AG, Waldenburg, Switzerland) were inserted by the same periodontist (T.T.Y.) in the present study. Pre-surgical radiographic evaluation was conducted using CBCT. Before surgery, the patient's mouth was rinsed with chlorhexidine mouthwash. After local anesthesia, full thickness flaps were reflected, and osteotomies were prepared in the first mandibular molar sites. In these surgical operations, 20 tissue-level and 20 bone-level dental implants 12 mm in length and 4.8 mm in diameter were inserted in Group I and Group II, respectively. Three months later, second-stage surgery was performed and implant exposed into the oral cavity. Cover screw was removed and replaced with healing abutments. Three months waited for second surgery in bone level implants. Patients of both groups were enrolled in a monthly periodontal/peri-implant maintenance program after abutments were connected in which, full mouth scaling was performed around all natural teeth and implant surfaces. Oral hygiene instructions regarding regular tooth brushing were given and patients were encouraged to floss the teeth and periimplant surfaces daily. There was no implant failed during the study and adverse event of these treatments.

ELIGIBILITY:
Inclusion Criteria:

* patients in the study who had one tooth absent in the mandible
* patients in the study should be least 18 years old.

Exclusion Criteria:

Patients in the study were the absence of the following points;

* poor mouth hygiene,
* bruxism, dental implants,
* chemotherapy or radiotherapy,
* addictions (alcohol, cigarettes, and medications),
* disease in the jawbones observed clinically or radiographically,
* pregnancy,
* antibiotic and/or anti-inflammatory medication use in the last three months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2010-10-01 (Actual); Study Completion 2011-06-01 (Actual)

PRIMARY OUTCOMES:
change of alveolar bone level | 0 and 6 month
  The primary outcome of the study was a change in alveolar bone level (height in mm) at the 40 implant site between T0 and T2 months after surgery measured on CBCT. All measurements were performed at four sites (mesial, distal, buccal, and lingual) around each dental implant at T0 and T2. These four values were then averaged for each dental implant.
  * Alveolar bone level were measured in millimeters (height in mm) from a fixed reference point on the implant (implant shoulder to the most coronal position of the crestal bone contacting the implant).

SECONDARY OUTCOMES:
changes level of IL-1β | 0, 3, and 6 month
  The secondary outcome of the study was change the level of IL-1β pg/ml between T0, T1, and T2. To obtain PICF, filter paper strips were gently inserted into the peri-implant crevice for 30 s at the mesial, distal, buccal, and lingual sites of the dental implant. A Williams periodontal probe was used for all clinical measurements.These parameters were recorded for evaluating the clinical status of the dental implants. All measurements were performed at four sites around each dental implant. For the statistical analysis, median of the four measurements at each implant was used.
  * The level of IL-1β pg/ml (weight in picogram, weight in milliliter)
changes of PPD | 0, 3, and 6 month
  The secondary outcome of the study was change of the PPD between T0, T1, and T2. A Williams periodontal probe was used for all clinical measurements.These parameters were recorded for evaluating the clinical status of the dental implants. All measurements were performed at four sites around each dental implant. For the statistical analysis, median of the four measurements at each implant was used.
  * Probing pocket depth (PPD) (depth in mm), were measured
changes of Modified plaque index | 0, 3, and 6 month
  The secondary outcome of the study was change of the Modified plaque index between T0, T1, and T2. A Williams periodontal probe was used for all clinical measurements.These parameters were recorded for evaluating the clinical status of the dental implants. All measurements were performed at four sites around each dental implant. For the statistical analysis, median of the four measurements at each implant was used.
  * Modified plaque index (0=no plaque, 1= mild plaque, 2= moderate plaque, 3=severe plaque).
changes of Modified gingival index | 0, 3, and 6 month
  The secondary outcome of the study was change of the Modified gingival index between T0, T1, and T2. A Williams periodontal probe was used for all clinical measurements.These parameters were recorded for evaluating the clinical status of the dental implants. All measurements were performed at four sites around each dental implant. For the statistical analysis, median of the four measurements at each implant was used.
  * Modified gingival index (0=healthy, 1=mild inflammation 2= moderate inflammation 3=severe inflammation).
changes of Modified bleeding index | 0, 3, and 6 month
  The secondary outcome of the study was change of the Modified bleeding index between T0, T1, and T2. A Williams periodontal probe was used for all clinical measurements.These parameters were recorded for evaluating the clinical status of the dental implants. All measurements were performed at four sites around each dental implant. For the statistical analysis, median of the four measurements at each implant was used.
  * Modified bleeding index (0= no bleeding, 1= mild bleeding, 2= moderate bleeding, 3=severe bleeding).

CONTACTS AND LOCATIONS:
Overall Officials: tuba talo yıldırım, Principal Investigator — Dicle University
Locations (1):
- Dicle University, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data can not be used another purpose such as meta-analyses, reanalysis, or replication of results.

REFERENCES:
- [Derived] Talo Yildirim T, Acun Kaya F, Yokus B, Colak M, Ozdemir Kaya E, Tekin G, Saribas E, Uysal E, Guncu GN. Associations of alveolar bone loss and interleukin-1beta levels in one- and two-stage surgical procedures: a randomized prospective trial. Acta Odontol Scand. 2017 Nov;75(8):608-615. doi: 10.1080/00016357.2017.1367959. Epub 2017 Aug 21. PMID 28826290
- Available data/document: Clinical Study Report — http://mc.manuscriptcentral.com/jperio